CLINICAL TRIAL: NCT04102254
Title: Thalamic Stimulation for Epilepsy Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lead acquisition from company & COVID-19 restrictions
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00103374
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Seizures; Epilepsy; Seizure Disorder
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ANT recording and stimulation (Experimental): Up to 15 adult patients who present to Duke Neurosurgery for routine seizure location using sEEG will be asked to enroll in this pilot study of ANT recording and stimulation. Once enrolled in the trial, subjects will have additional placement of two thalamic electrodes during the course of standard sEEG placement surgery. Patients routinely remain hospitalized for 7-14 days after sEEG placement, during which time their seizure medications are tapered. Continuous neural recordings are made through the sEEG electrodes for the purposes of seizure localization during the entire time the depth electrodes are in place. Up to three times daily, standard intermittent high-frequency stimulation [130 Hertz (Hz), 90-millisecond pulse width, and 2 milliamps (mA) intensity] will be performed with a 60-seconds on and a 300-seconds off cycle following surgery up to the entire length of sEEG monitoring.
  Interventions: Procedure: ANT recording and stimulation

INTERVENTIONS:
Procedure: ANT recording and stimulation — In this study, the investigator aims to perform sEEG recordings during simultaneous ANT recording and stimulation to better understand the following: 1) how the ANT is involved in various seizure types; 2) which cortical regions are modulated by established ANT stimulation patterns; and 3) how novel ANT stimulation patterns modify epileptogenic cortical activity.

SUMMARY:
In this study, the investigator aims to perform cortical stereo electroencephalogram (sEEG) recordings during simultaneous anterior nucleus of the thalamus (ANT) recording and stimulation to better understand the following: 1) how the ANT is involved in various seizure types; 2) which cortical regions are modulated by established ANT stimulation patterns; and 3) how novel ANT stimulation patterns modify epileptogenic cortical activity. Together, this knowledge will advance ANT deep brain stimulation (DBS) therapy by providing a physiologic basis for patient selection for ANT DBS, while identifying brain signals and stimulation patterns that can be used to develop novel methods for ANT DBS. Up to 15 adult patients (18 and older) who present to Duke Neurosurgery for routine seizure localization using sEEG will be asked to enroll in this pilot study of ANT recording and stimulation. In the course of surgical epilepsy treatment, patients routinely undergo surgical placement of sEEG electrodes for the purposes of seizure localization. During this procedure, 2 additional leads will be placed in the ANT. These patients remain hospitalized for 7-14 days after sEEG placement, during which time their seizure medications are tapered. Concurrent video monitoring is performed while continuous neural recordings are made through the sEEG electrodes. Additionally, continuous recordings will be performed through the electrodes placed in the thalamus. Periodically, standard intermittent high-frequency stimulation (130 Hz, 90-ms pulse width, and 2 mA intensity) will be performed with a 60-s on and a 300-s off cycle after surgery. These standard ANT stimulation parameters are employed clinically. Data will include the sEEG recordings marked for ANT stimulation, any side effects, medications, past medical history (PMH), and tests/procedures during the hospital stay. Risks involved are as described for the standard depth electrode surgery with the addition of the possible side effects from the stimulation which include sensations of numbness and tingling, and possibly increased seizure activity.

DETAILED DESCRIPTION:
The purpose of this research is to examine the physiologic underpinnings of deep brain stimulation of the anterior nucleus of the thalamus (ANT), a method reducing seizures in adults diagnosed with medically refractory epilepsy. In this study, the investigator aims to perform cortical stereo electroencephalogram (sEEG) recordings during simultaneous ANT recording and stimulation to better understand the following: 1) how the ANT is involved in various seizure types; 2) which cortical regions are modulated by established ANT stimulation patterns; and 3) how novel ANT stimulation patterns modify epileptogenic cortical activity. Together, this knowledge will advance ANT DBS therapy by providing a physiologic basis for patient selection for ANT DBS, while identifying brain signals and stimulation patterns that can be used to develop novel methods for ANT DBS.

Approximately 3 million people in the United States experience epilepsy. Despite medical therapy, up to 30% of these patients continue to experience recurrent seizures. In this medically refractory population, tissue resection or ablation offer a high likelihood of seizure freedom, if a single epileptogenic focus can be precisely identified. For patients who are not candidates for resection or ablation, or those who continue to have seizures after these treatments, neuromodulation represents an alternative therapeutic option. One such therapy, deep brain stimulation (DBS) has been approved for around 5 years in Europe and was recently approved in the United States as a treatment for medically refractory epilepsy.

A number of potential DBS targets are being investigated, particularly, the ANT, which consists of the anteroventral, anterodorsal, and anteromedial nuclei. The ANT was recognized as a potential target because of its central connectivity to cortical regions where seizures often originate. Several pilot studies and recent trials have demonstrated 5-year efficacy and safety outcomes for ANT DBS. In a large randomized controlled study of ANT stimulation with long-term follow-up, there was a 56% median seizure reduction at the 2 year, and a 69% median and seizure reduction at the 5 year, in patients with drug-resistant focal epilepsy. This study also suggested that patients with temporal lobe epilepsy achieved greater benefit than those with extra-temporal or multifocal seizures. Since these pivotal trials, DBS of the ANT has emerged as a promising therapy for focal drug resistant epilepsy, however, its basic mechanism of action is unclear. One study which examined cortical local field potentials recordings during high-frequency ANT stimulation (130 Hz), has suggested that epileptic network desynchronization is a potential mechanism of DBS of the ANT.

ELIGIBILITY:
All epilepsy patients admitted to Duke Hospital for surgical placement of depth electrodes age 18 and up are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-07 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Percent changes from baseline in power (dB) | Measurements will be made 7-14 days following surgery for sEEG placement
  Differences of greater than 25% in magnitude in percent mean change in power between primary regions of interest will be reported. A maximum of 20 comparisons will be made.
Percent changes from baseline in rates of interictal spikes | Measurements will be made 7-14 days following surgery for sEEG placement
  Differences of greater than 25% in magnitude in percent mean change in rates of interictal spikes between primary regions of interest will be reported. A maximum of 20 comparisons will be made.
Percent changes from baseline in rates of high frequency oscillations | Measurements will be made 7-14 days following surgery for sEEG placement
  Differences of greater than 25% in magnitude in percent mean change in rates of high frequency oscillations between primary regions of interest will be reported. A maximum of 20 comparisons will be made.
Percent changes in connectivity density | Measurements will be made 7-14 days following surgery for sEEG placement
  Changes of greater than 25% in magnitude in connectivity density on versus off stimulation in primary regions of interest will be reported. A maximum of 20 comparisons will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Southwell, M.D., Ph.D., Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Study data will be stored in the Duke Research Electronic Data Capture (REDCap) database.